CLINICAL TRIAL: NCT07053332
Title: A Single-arm, Prospective Phase II Clinical Study of Neoadjuvant PD-1/CTLA-4 Combination Antibody With Low-dose Radiotherapy in Resectable dMMR/MSI-H Esophagogastric Junction/Gastric Adenocarcinoma.
Brief Title: A Study on Immunotherapy Combined With Radiotherapy for Esophagogastric Junction/Gastric Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, Chao Yue, Chief Physician, Jiangsu Cancer Institute & Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: neoCACR for dMMR/MSI-H G/GEJ
Record Dates: First submitted 2025-06-15; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Esophagogastric Junction/Gastric Adenocarcinoma
Keywords: Iparomlimab and Tuvonralimab，Radiotherapy，esophagogastric junction/gastric adenocarcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1/CTLA-4 combination antibody with low-dose radiotherapy (Experimental)
  Interventions: Drug: PD-1/CTLA-4 combination antibody with low-dose radiotherapy

INTERVENTIONS:
Drug: PD-1/CTLA-4 combination antibody with low-dose radiotherapy — * PD-1/CTLA-4 combination antibody: Iparomlimab and Tuvonralimab， 5mg/kg on day 1, day 22, and day 43, administered via intravenous infusion, for a total of three cycles before surgery and maintained for up to 1 year after surgery.
  * Radiotherapy: To be conducted within one week of the start of immunotherapy, with a total dose of DT: 30Gy, 2.5Gy × 12 fractions, once daily, five times per week. The preoperative radiotherapy target area will be delineated by the radiation oncologist in accordance with the "NCCN Guidelines for Gastric/Esophagogastric Junction Cancers 2022" and in consultation with the opinions of the general surgeon.
  * Surgery: Surgical treatment will be completed within 3-5 weeks after the completion of neoadjuvant therapy.
  * Adjuvant therapy: Postoperative immunotherapy will be maintained for up to 1 year.

SUMMARY:
A single-arm, prospective phase II clinical study of neoadjuvant PD-1/CTLA-4 combination antibody with low-dose radiotherapy in resectable dMMR/MSI-H esophagogastric junction/gastric adenocarcinoma.

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-arm Phase II clinical trial. Participants will be patients with resectable locally advanced dMMR/MSI-H esophagogastric junction/gastric adenocarcinoma staged as cT1-2N1-3M0 or T3-T4aN0-3M0 according to the AJCC/UICC staging system. The objective of this study is to evaluate the safety and efficacy of PD-1/CTLA-4 combination antibody therapy combined with low-dose radiotherapy in patients with locally advanced resectable dMMR/MSI-H esophagogastric junction/gastric adenocarcinoma.

Eligible participants who meet the inclusion criteria will be enrolled in the study.

Primary endpoint: Pathological complete response rate (pCR), defined as pT0N0M0，Safety: Treatment-related adverse reactions of grade 3 or above according to CTCAE 5.0 will be recorded from the start of treatment until 30 days after surgery..

Secondary endpoints:

Treatment feasibility: the proportion of patients who complete neoadjuvant therapy and undergo surgery within 3-5 weeks after treatment.

Major pathological response rate (MPR): the percentage of residual viable tumor cells in the tumor bed after neoadjuvant therapy ≤10%.

Imaging-assessed response rate: evaluated using multimodal imaging including CT/GI ultrasound and MRI.

R0 resection rate: the proportion of patients achieving R0 resection among all enrolled patients.

Treatment safety: recorded using CTCAE 5.0 for grade 3 or higher treatment-related adverse events, from the start of neoadjuvant therapy until 30 days after surgery.

Postoperative complications: assessed using the Clavien-Dindo classification. Time to recurrence (TTR): time from the start of the study to the first documented recurrence.

Progression-free survival (PFS): time from the start of the study to tumor progression (in any aspect) or death from any cause.

Overall survival (OS): time from the start of the study to death from any cause.

Treatment schedule:

The maximum interval between participant screening and initiation of treatment is 3 weeks (≤21 days).

PD-1/CTLA-4 combination antibody: Eparaplimab Icotinib Injection, 5 mg/kg on Day 1, Day 22, and Day 43, administered intravenously, for a total of three cycles.

Radiotherapy: Initiated within one week of starting immunotherapy, total dose DT: 30 Gy, 2.5 Gy × 12 fractions, once daily, five times per week.

Surgery: Performed 3-5 weeks after completion of neoadjuvant therapy. Postoperative adjuvant therapy: Eparaplimab Icotinib Injection, 5 mg/kg on Day 1, every 3 weeks (Q3W), administered intravenously, continued up to 1 year.

The study continues until disease progression, voluntary withdrawal by the patient, or occurrence of intolerable toxicities. Efficacy and safety assessments are conducted every two cycles (42 days ±7 days). If disease progression is observed (based on investigator evaluation or imaging evidence), the patient will voluntarily withdraw from the study; if intolerable toxicities occur, the participant should discontinue study treatment. In the event of treatment discontinuation for any reason, a final study visit should be conducted approximately 12 weeks after the last dose of study drug, to collect all possible adverse events and concomitant medication information. Follow-up of drug-related or possibly related adverse events should continue until the event stabilizes or resolves.

A notice of study completion will be submitted to the hospital's Clinical Trial Management Center based on the date of the final follow-up visit of the last enrolled participant. An update and status annotation will also be made at the clinical trial registry.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study, sign the informed consent form, demonstrate good compliance, and agree to follow-up;
2. Patients with esophagogastric junction/gastric adenocarcinoma (Siewert type II/III) confirmed by endoscopic pathology (note: pathologies from other hospitals must be reviewed at our hospital), with dMMR/MSI-H status confirmed by immunohistochemistry or genetic testing;
3. Based on endoscopic, CT, MRI, or PET-CT findings, AJCC 8th edition staging is cT1-2N1-3M0 or T3-T4aN0-3M0;
4. Age between 18 and 80 years, inclusive of both 18 and 80, both genders are eligible;
5. ECOG PS score of 0-1;
6. Presence of measurable and/or non-measurable lesions as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1);
7. No prior systemic anti-tumor treatment (including but not limited to systemic chemotherapy, radiotherapy, molecular targeted therapy, immunotherapy, biologic therapy, local therapy, or investigational drugs);
8. The function of major organs must meet the following criteria (no blood components or cell growth factors allowed within 2 weeks before screening):

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
   * Platelets ≥ 100 × 10⁹/L;
   * Hemoglobin ≥ 9 g/dL;
   * Serum albumin ≥ 2.8 g/dL;
   * Total bilirubin ≤ 1.5 × ULN, ALT, AST, and/or ALP ≤ 2.5 × ULN;
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula);
   * International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN (patients receiving stable-dose anticoagulation therapy such as low-molecular-weight heparin or warfarin with INR within the expected therapeutic range may be enrolled).

Females of childbearing potential should undergo a urine or serum pregnancy test within 72 hours prior to the first dose of study drug and must have a negative result. They must also agree to use effective contraception during the study period and for 5 months after the last dose. Male participants whose partners are of childbearing potential must also use effective contraception during the study period and for 7 months after the last dose.

Exclusion Criteria:

1. History of surgery for gastric or gastroesophageal junction tumor;
2. Immunohistochemistry or genetic testing shows pMMR, MSI-L, or MSS;
3. High risk of gastrointestinal bleeding or perforation;
4. Poor nutritional status, BMI < 18.5 kg/m², or PG-SGA score ≥ 9;
5. Major surgery or serious trauma within 4 weeks prior to the first use of the study drug;
6. Presence of uncontrollable pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
7. Previously received or is currently receiving any of the following treatments: anti-PD-1 or anti-PD-L1 antibody therapy, chemotherapy, radiotherapy, targeted therapy;
8. Received any investigational drug within 4 weeks prior to the first use of the study drug;
9. Requires systemic corticosteroids (more than 10 mg/day prednisone equivalent) or other immunosuppressive agents within 2 weeks prior to the first use of the study drug, except for local inflammation of the esophagus/stomach and corticosteroid use for allergy prevention or nausea/vomiting control. Special circumstances require communication with the sponsor. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal corticosteroid replacement at doses >10 mg/day prednisone equivalent are allowed;
10. Has received an anticancer vaccine or received a live vaccine within 4 weeks prior to the first administration of the study drug;
11. Has any active autoimmune disease or history of autoimmune disease (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism), except for vitiligo or resolved childhood asthma/allergy that does not require intervention in adulthood. Patients on stable-dose thyroid hormone replacement for autoimmune hypothyroidism and those on stable-dose insulin for type I diabetes mellitus may be included;
12. History of immunodeficiency, including HIV-positive status, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation or allogeneic bone marrow transplantation;
13. Any condition requiring systemic corticosteroid treatment (higher than 10 mg/day prednisone or equivalent) or other immunosuppressive therapy within 14 days before treatment initiation (except for the following situations: locally applied, ophthalmic, intra-articular, intranasal, or inhaled corticosteroids with minimal systemic absorption; short-term (≤7 days) prophylactic use of corticosteroids (e.g., for contrast agent allergy prevention) or for non-autoimmune conditions (e.g., delayed hypersensitivity reactions due to allergen exposure));
14. Presence of uncontrolled cardiac symptoms or diseases such as (1) NYHA class II or higher heart failure, (2) unstable angina, (3) myocardial infarction within 1 year, or (4) clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
15. Severe infection (CTCAE > Grade 2) within 4 weeks prior to the first use of the study drug, such as severe pneumonia requiring hospitalization, bacteremia, or infectious complications; baseline chest imaging suggests active pulmonary infection; signs or symptoms of infection requiring oral or intravenous antibiotic treatment within 2 weeks prior to enrollment, except for prophylactic antibiotic use;
16. History of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, or other uncontrolled acute pulmonary diseases;
17. Evidence of active tuberculosis infection by medical history or CT findings, or history of active tuberculosis within 1 year prior to enrollment, or history of active tuberculosis more than 1 year ago without proper treatment;
18. Active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10⁴ copies/mL) or hepatitis C (anti-HCV positive and HCV-RNA above the lower limit of detection of the assay method);
19. Laboratory abnormalities in sodium, potassium, or calcium levels greater than Grade 1 within 2 weeks prior to enrollment, which cannot be corrected after treatment;
20. Known allergy, hypersensitivity, or contraindication to macromolecular protein preparations, PD-1 components, paclitaxel, capecitabine, or any excipients in their formulations;
21. History of any other malignancy, except for low-risk malignancies with low metastasis and mortality risk (5-year survival rate >90%), such as adequately treated basal cell or squamous cell skin cancer or cervical carcinoma in situ;
22. Pregnant or lactating women; fertile subjects unwilling or unable to take effective contraceptive measures;
23. The investigator determines that the subject has other factors likely to result in premature termination of the study, such as other serious illnesses (including mental illness) requiring concurrent treatment, recent serious illnesses (e.g., myocardial infarction, cerebrovascular accident) with high recurrence risk, severely abnormal laboratory values, family or social factors that may affect the subject's safety or data collection from the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-08-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | Assessed average of 1 month after surgery
  Pathological complete response is defined as pT0N0M0.
Safety | From the start of treatment until 30 days after surgery
  Treatment-related adverse reactions of grade 3 or above according to CTCAE 5.0 will be recorded from the start of treatment until 30 days after surgery.

SECONDARY OUTCOMES:
Major pathological response rate (Major pathological response, MPR) | Assessed average of 1 month after surgery
  After neoadjuvant therapy, the percentage of residual viable tumor cells within the tumor bed is ≤10%.
R0 resection rate (Complete Resection With no Tumor Within 1 mm of the Resection Margins (R0) Rate) | Assessed average of 1 month after surgery
  The proportion of patients who achieve R0 resection among all enrolled patients.
Post-operative complications | Assessed average of 1 month after surgery
  Assessed using the Clavien-Dindo classification
Time to relapse (Time to Relapse, TTR) | From the time of enrollment, until the disease relapses or metastasizes，assessed up to 5 years follow-up.
  The time from the start of the study to the first documented relapse.
Progression-free survival (Progression-free survival, PFS) | From the time of enrollment, until the disease relapses or metastasizes，assessed up to 5 years follow-up.
  The time from the start of the study to tumor progression (in any aspect) or death (from any cause).
Overall survival (Overall Survival, OS) | From the time of enrollment, until the disease relapses or metastasizes，assessed up to 5 years follow-up.
  The time from the start of the study to death from any cause.

IPD SHARING:
Plan to Share IPD: No